CLINICAL TRIAL: NCT01299974
Title: Project PARIS: Parents and Residents in Session
Acronym: PARIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Picker Institute (Unknown); The Arnold P. Gold Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 10-1621
Record Dates: First submitted 2011-02-08; First posted 2011-02-21 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Family-centered Care
Keywords: Family-centered; teaching; residents; family faculty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parents and Residents in Session (Other): Parents and Residents in Session
  Interventions: Other: Parents and Residents in Session

INTERVENTIONS:
Other: Parents and Residents in Session — Family Faculty members agreed to participate in meetings with pediatric residents who agree to participate. Standardized meetings include discussions of the following: 1. Impact of hospitalization on the behavior and development of each participating parent's child. 2. Effective communication with a parent 3. How to gain trust 4. The family meeting: who participates, the agenda 5. Troubleshooting: how to deal with difficult situations (the parents will present a few instances, from their own experience, which they think might be challenging to the clinicians who treated their children). Other core components will be added (or existing ones deleted) based on participants' feedback. The meeting will be attended by two residents, a family council member, and a senior faculty who will serve as monitor. Following the meeting, the residents will have an opportunity to ask questions and offer comments about the experience in a dedicated feedback interview with a senior faculty member.
  Other Names: Parents and Residents in Session to improve family-centered care

SUMMARY:
The study seeks to implement and test a novel approach to teach pediatric residents about patient and family-centered care (PFCC). The approach calls for a supervised meeting between a family member of a previously hospitalized child and a resident in the context of a pediatric residency rotation.

DETAILED DESCRIPTION:
A specific patient and family centered care module will be implemented in the context of an existing training rotation. This module includes a meeting between resident physicians (trainees) and parents of previously hospitalized children (members of the Family Faculty in our institution), monitored by a senior faculty member. Patient and family centered care will be discussed using predefined, manual-driven guidance. This meeting is followed by a discussion with the faculty member to identify core components of family-centered care as exemplified in the parent interview.

ELIGIBILITY:
Inclusion Criteria:

* Residents in good standing in a pediatric residency at Mount Sinai Medical
* Center who agree to participate in the study

Exclusion Criteria:

* Residents who did not agree to participate
* Residents who have less than 3 months to complete their residency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Resident's knowledge | The difference between values obtained at baseline (upon recruitment) and values obtained within 24 hours after completion of the interview
  Residents' knowledge about family-centered care as measured by a questionnaire

SECONDARY OUTCOMES:
Residents' attitude towards family-centered care as measured by a questionnaire | The difference between values obtained at baseline (upon recruitment) and values obtained within 24 hours after completion of the interview
Parents' acceptance of family-centered care as measured by a questionnaire | The difference between values obtained at baseline (upon recruitment) and values obtained within 24 hours after completion of the interview

CONTACTS AND LOCATIONS:
Overall Officials: Joel Forman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Kravis Children's Hospital, New York, New York, United States